CLINICAL TRIAL: NCT07287865
Title: Study Title: Oncological and Functional Results After Total Laryngectomy and Pharyngolaryngectomy
Acronym: TL&TPL
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Marco Benazzo, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: TL&TPL
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-01

CONDITIONS: Laryngeal and Hypopharyngeal Tumors
MeSH Terms: conditions — Laryngeal Diseases | interventions — Surgical Flaps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- reconstructive flap: patients affected by laryngeal and/or hypopharyngeal carcinoma who underwent/undergo total laryngectomy, total hemipharyngolaryngectomy, or circular pharyngolaryngectomy, with reconstructive flap, from January 2015 to December 2030
  Interventions: Procedure: surgical flap
- NO reconstructive flap: patients affected by laryngeal and/or hypopharyngeal carcinoma who underwent/undergo total laryngectomy, total hemipharyngolaryngectomy, or circular pharyngolaryngectomy,without reconstructive flap, from January 2015 to December 2030

INTERVENTIONS:
Procedure: surgical flap — Pedicled or free flap was harvested and placed over the pharyngeal suture (on-lay) following TL or tunnelled to reconstruct wide defects (in-lay) after TPL.
  Groups: reconstructive flap

SUMMARY:
Salvage total laryngectomy (TL) and total pharyngolaryngectomy (TPL) are the gold standard for most recurrent laryngeal and hypopharyngeal tumors as well as in patients with contraindication for chemoradiotherapy (CRT). Free or pedicled flaps are the two mandatory options for pharyngeal reconstruction after TPL, while remain an optional indication to protect the neopharynx after TL. The most common complication after TL or TPL is pharyngocutaneous fistula (PCF), with an incidence ranging from 3% to 65%, according to the surgical defect and type of reconstruction. The etiology of PCF is multifactorial and the most important risk factors are a history of CRT, low hemoglobin levels (< 12.5 g/dl), and malnutrition. A growing concern is the role of nutritional status, with sarcopenia as an emergent risk factor for post-operative complications, because muscle wasting negatively influences wound healing and overall recovery. Salivary stent placement, 3-layers neopharyngeal sutures, cricopharyngeal myotomy and prophylactic use of vascularized flaps are possible protective factors to reduce the risk of PCF. Despite these evidences, it remains unclear which are the best candidates for flap reconstruction, as well as which preoperative risk factors influence the risk of PCF.

The rationale of this ambispective monocentric study is to identify the risk factors statistically significant associated with the development of PCF and the influence of preoperative sarcopenia on postoperative complications risks following TL and TPL.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing to TL with direct closure of the pharynx or TPL and reconstruction of the pharynx with a free or pedicled flap in cases of:

* Naive laryngeal neoplasia (cT1-cT4a with possible extension to the esophagus, oropharynx, or hypopharynx);
* Recurrence of laryngeal or hypopharyngeal cancer in patients previously treated with surgical intervention (TLM/CO2 laser or OPHL);
* Recurrence of laryngeal or hypopharyngeal cancer in patients previously treated with RT or CRT;
* Loss of laryngeal function induced by RT, CRT, or OPHL treatment;
* Availability of data according to the assessments that must be made, including a follow-up period of at least 2 months.

Exclusion Criteria:

* Lack of useful data to carry out the assessments related to the study itself

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by laryngeal and/or hypopharyngeal carcinoma who underwent/undergo total laryngectomy, total hemipharyngolaryngectomy, or circular pharyngolaryngectomy, with or without reconstructive flap, at Fondazione IRCCS Policlinico San Matteo from January 2015 to December 2030
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The association between the use of a surgical flap and the incidence of post-operative fistulas during follow-up | within 30 days from surgery
  Proportion of subjects who develop a post-operative fistula (blind or pharyngo-cutaneous fistula, PCF, with or without the use of a surgical flap, which develop within 30 days from surgery

SECONDARY OUTCOMES:
The association between the use of a surgical flap and the incidence of mid to longterm post-operative fistulas | 30 days and at mid to long term.
  The rate of development of a mid to longterm post-operative fistula
Potential correlates of fistulas development both within 30 days and at mid to long term | 30 days and 36 months
  * Demographic and medical history
  * Tumor characteristics
  * Previous tumor treatment
  * Laboratory
  * Perioperative management
The incidence of any post-operative complications | 1-36 months follow-up
  Fistulas and any of the surgical and non surgical complications within 30 days.
  Surgical complications (require reintervention):
  * Necroses
  * Hematoma/hemorrage
  * Neopharyngeal stenosis
  Non surgical Complications:
  * Hypocalcemia
  * Anemia requiring blood transfusion
  * Hypokalemia
  * Pneumonia
  * Cardiac complications
  * Infection
36 months incidence of tumor related events | 36 months after surgery
  Potential correlates will be:
  * The combination of surgical flap and fistula
  * The lymphnode ratio </≥18 (LNR, calculated as the number of positive lymph nodes divided by the total number of lymph nodes removed, including both positive and negative nodes )
  * Sarcopenia
The prognostic role of both the use of a surgical flap and the development of post-operative fistulas | 36 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marco Benazzo, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (1):
- SC Otorinolaringoiatria - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No